CLINICAL TRIAL: NCT02387905
Title: Prophylactic Cement Augmentation for Patients at High Risk for Developing Vertebral Body Compression Fracture Following Spine Stereotactic Radiosurgery: A Randomized Phase II Clinical Trial
Brief Title: Cement Augmentation in Preventing Vertebral Body Compression Fracture Following Spine Stereotactic Radiosurgery in Patients With Solid Tumors and Spinal Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0561; NCI-2015-00494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0561 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignant Neoplasm in the Spine; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients undergo stereotactic spinal radiosurgery per standard of care.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery
- Arm II (vertebral body cement augmentation) (Experimental): Patients undergo vertebral body cement augmentation within 4 weeks before or after standard stereotactic spinal radiosurgery.
  Interventions: Procedure: Management of Therapy Complications; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Management of Therapy Complications — Undergo vertebral body cement augmentation
  Arms: Arm II (vertebral body cement augmentation)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo standard stereotactic spinal radiosurgery
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This randomized phase II trial studies how well cement augmentation works in preventing vertebral body compression fracture following spine stereotactic radiosurgery in patients with solid tumors that have spread to the spine. Spine stereotactic radiosurgery delivers a high dose of radiation to vertebral metastases and can sometimes lead to a vertebral compression fracture. Using body cement on the largest part of the vertebra (a procedure called vertebral body cement augmentation) may help prevent a fracture after stereotactic spinal radiosurgery. It may also lessen pain and improve quality of life in patients with solid tumors and spinal metastases undergoing this surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether prophylactic cement augmentation reduces new or progressive vertebral body fracture at 3 months in high risk patients undergoing single fraction spine stereotactic radiosurgery.

SECONDARY OBJECTIVES:

I. To assess the impact of prophylactic cement augmentation on time to first new or progressive vertebral body fracture.

II. To assess the impact of prophylactic cement augmentation on pain control measured every three months post treatment.

III. To assess the impact of prophylactic cement augmentation on quality of life measured every three months post treatment.

IV. To estimate local control in each arm. V. To estimate overall survival in each arm. VI. To document and assess post-treatment adverse side effects between the two arms.

VI. To document and assess the relationship between radiographic vertebral body fracture, pain control and quality of life.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo stereotactic spinal radiosurgery per standard of care.

ARM II: Patients undergo vertebral body cement augmentation within 4 weeks before or after standard stereotactic spinal radiosurgery.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologic proof of solid tumor malignancy and radiographic evidence of spine metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* All patients must be able to lie supine
* All patients must have no more than 3 contiguous vertebral body levels treated at a single site, and no more than 3 discontiguous vertebral body levels treated
* All patients must have a single fraction spine radiosurgery at the designated site of interest to at least a dose of 18 Gray (Gy)
* All patients must be deemed at "high risk" of developing vertebral body fracture by having at least one of the following characteristics:

  * Spine Instability Neoplastic Score classification of "Indeterminate" deemed as a score from 7 to 12
  * Pre-existing vertebral body fracture
  * Planned radiation dose of 24 Gy
* All patients must have a vertebral body site to be treated located from T1 to L5
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* All patients must sign informed consent verifying that they are aware of the investigational nature of this study in keeping with the rules and policies of M.D. Anderson Cancer Center; the only acceptable consent is the one approved by M.D. Anderson Institutional Review Board (IRB)
* Patients undergoing bisphosphonate therapy are allowed

Exclusion Criteria:

* Patients who have had prior radiotherapy at the spine site and level to be treated
* Patients who have had prior surgery at the spine level to be treated to include prior cement augmentation, laminectomy, vertebrectomy, tumor debulking, instrumentation
* Patients with gross disease involving only the posterior elements
* Patients who have > 50% vertebral body collapse
* Patients unable to undergo magnetic resonance imaging (MRI) of the spine
* Patents with cord compression
* Patients deemed not be a candidate for cement augmentation for any reason
* Patients who have frank mechanical pain
* Patients with both pedicles involved with gross disease at the level of potential cement augmentation
* Pregnant women are excluded from this study
* Patients with a histology of lymphoma, myeloma and small cell lung cancer histologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vertebral compression fracture rate | At 3 months
  Will compare the 3-month vertebral compression fracture proportions between treatment groups using the Fisher exact test. Will be performed on the intention-to-treat principle.

SECONDARY OUTCOMES:
Time to first new or progressive vertebral body fracture | Up to 2 years
  To assess the impact of prophylactic cement augmentation on time to first new or progressive vertebral body fracture, will use the Kaplan-Meier method to estimate the freedom from fracture curves and Cox proportional hazards regression analysis to estimate the hazard ratio with confidence intervals and associated p-values.
Pain control, assessed using the Brief Pain Inventory form | Up to 2 years
  Will use mixed effects linear models to analyze this longitudinal data.
Quality of life, assessed using the MD Anderson Symptom Inventory-Spine Tumor form | Up to 2 years
  Participants are asked to recall symptom severity and interference during the past 24 hours. Part I, The severity of the symptoms, including pain, fatigue, nausea, disturbed sleep, short of breath etc. Part II, How have the symptoms interfered with patient life, including mood, work, relations with other people etc. Part I, range 0-10. A score of 0 would mean the symptom is not present and a score of 10 means the symptom is as bad as you can imagine). Part II, range 0-10 (A score of 0 would mean the symptom did not interfere; A score of 10 means the symptom has interfered completely. The ratings in the MDASI can be averaged into several subscale scores: mean core symptom severity, mean module symptom severity, mean total symptom severity, and mean interference. The interference items can further be broken down into mean activity interference and mean affective interference. Symptom items may be presented individually
Local control | Up to 2 years
  Will estimate time to first local failure curves using the Kaplan-Meier method.
Overall survival | Up to 2 years
  Will use the Kaplan-Meier method.
Incidence of post-treatment adverse events | Up to 2 years
  Will estimate the difference in grade 3+ toxicity rates, with 95% confidence intervals and a chi-squared test p-value.
Radiographic vertebral body fracture, pain control and quality of life assessment | Up to 2 years
  Will assess the relationship between radiographic vertebral body fracture, pain control and quality of life using correlation analyses. Additional analyses may be conducted as appropriate.
Quality of life, assessed using the EuroQol 5-dimensional 5-level questionnaire. | Up to 2 years
  Will use mixed effects linear models to analyze this longitudinal data. The questionnaire consists 2 parts.
  Part 1 is descriptive system (participants are asked mobility, self-care status, usual activities, pain/discomfort, anxiety/depression, and each dimension has 5 levels;
  Part 2 is the Visual analogue scale (the self-rated health today with score 0-100; 100 means the best health you can imagine. 0 means the worst health you can imagine) Part 2, participants give self-rated health today with 100 means the best health you can imagine. 0 means the worst health you can imagine. Part 2, higher range represents a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amol J Ghia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org